CLINICAL TRIAL: NCT00485303
Title: A Phase II Open Label Study of CB7630 (Abiraterone Acetate) and Prednisone in Patients With Advanced Prostate Cancer Who Have Failed Androgen Deprivation and Docetaxel-Based Chemotherapy
Brief Title: An Efficacy and Safety Study of Abiraterone Acetate and Prednisone in Participants With Prostate Cancer Who Failed Androgen Deprivation and Docetaxel-Based Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cougar Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016921; COU-AA-004; 2007-002725-74 (EudraCT Number)
Record Dates: First submitted 2007-06-08; First posted 2007-06-12 (Estimated); Results first posted 2013-06-17 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Prostatic Neoplasms; Prostate Cancer
Keywords: Prostatic Neoplasms; Prostate cancer; Abiraterone acetate; CB7630; Prednisone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abiraterone (Experimental): Abiraterone acetate 1000 milligram (mg) (4 oral tablets of 250 mg each) will be administered once daily along with 5 mg oral prednisolone tablet administered twice daily for 28-days dosing cycle and will be continued until disease progression or unacceptable toxicity.
  Interventions: Drug: Abiraterone acetate; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone acetate — Abiraterone acetate oral tablets 250 milligram (mg) each will be administered at a total dose of 1000 mg until documented disease progression or unacceptable toxicity.
Drug: Prednisone — Prednisone/Prednisolone 5 mg tablet will be taken orally twice daily.
  Other Names: CB7630

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of abiraterone acetate in participants with advanced prostate cancer (a disease in which cells in the prostate gland become abnormal and start to grow uncontrollably, forming tumors).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single-arm, multicenter (when more than one hospital or medical school team work on a medical research study) study to evaluate the anti-tumor activities and safety of abiraterone acetate in participants with prostate cancer who have failed androgen deprivation and docetaxel-based chemotherapy. Abiraterone acetate oral tablet will be administered as a total dose of 1000 milligram (mg) orally (by mouth) once daily after an overnight fast and prednisone/prednisolone will be administered as 5 mg oral tablet twice daily. Participants will be enrolled and treated up to 12 cycles (or longer, if they have not progressed and continue to benefit from treatment). The study will consist of 3 parts: Screening (14 days), Open-label Treatment; and follow-up (up to 60 months). Participants will be evaluated primarily for prostate specific antigen response according to Prostate Specific Antigen Working Group (PSAWG) criteria. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma (malignant epithelial tumor with a glandular organization)of the prostate (a gland in the male reproductive system found below the bladder and in front of the rectum), but not with neuroendocrine (specialized neurons that produce hormones, such as neuropeptides or biogenic amines) differentiation or of small cell histology
* Prior chemotherapy (treatment of disease, usually cancer, by chemical agents) for prostate cancer with regimen(s) containing docetaxel
* Documented prostate specific antigen (PSA) progression according to Prostate Specific Antigen Working Group (PSAWG) eligibility criteria with a PSA more than (>) 5 nanogram per milliliter (ng/mL) or objective progression by Response Evaluation Criteria in Solid Tumors (RESIST) criteria
* Ongoing androgen deprivation with serum testosterone less than (<) 50 nanogram per deciliter (ng/dL)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of less than equal to (<=) 2 (Karnofsky Performance Status >= 50 percent)

Exclusion Criteria:

* Active or uncontrolled autoimmune disease (disorder in which a person's immune system attacks parts of his or her own body) that may require corticosteroid therapy
* Serious or uncontrolled co-existent non-malignant disease, including active and uncontrolled infection
* Uncontrolled hypertension (high blood pressure)
* Hemoglobin <=9.0 gram per deciliter (g/dL) without growth factor or transfusion support
* Abnormal liver (large organ that helps in many body functions, including digestion, metabolism, and storage of substances) function

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cougar Biotechnology, Inc. Clinical Trial, Study Director — Cougar Biotechnology, Inc.
Locations (14):
- United States (12):
  - UCLA, Los Angeles, California
  - Los Angeles, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - San Francisco, California
  - John Hopkins, Baltimore, Maryland
  - Baltimore, Maryland
  - Masachussetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Hospital, Boston, Massachusetts
  - Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York, New York
- United Kingdom (2):
  - Royal Marsden Hospital, Sutton
  - Sutton

REFERENCES:
- [Derived] Danila DC, Anand A, Sung CC, Heller G, Leversha MA, Cao L, Lilja H, Molina A, Sawyers CL, Fleisher M, Scher HI. TMPRSS2-ERG status in circulating tumor cells as a predictive biomarker of sensitivity in castration-resistant prostate cancer patients treated with abiraterone acetate. Eur Urol. 2011 Nov;60(5):897-904. doi: 10.1016/j.eururo.2011.07.011. Epub 2011 Jul 14. PMID 21802835
- See also: NATIONAL CANCER INSTITUTE — http://www.cancer.gov/
- See also: PROSTATE CANCER — http://www.nlm.nih.gov/medlineplus/prostatecancer.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Abiraterone: Abiraterone acetate 1000 milligram (mg) (4 oral tablets of 250 mg each) was administered once daily along with 5 mg oral prednisolone or prednisone tablet administered twice daily for 28-days dosing cycle and was continued until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Abiraterone
Started | 58
Completed | 2
Not Completed | 56
Not completed — Adverse Event | 5
Not completed — Progressive Disease | 44
Not completed — Other | 3
Not completed — Initiation of new anti-cancer treatment | 2
Not completed — Treatment ongoing at cutoff date | 2

BASELINE CHARACTERISTICS:
Arm/Group | Abiraterone
Number analyzed (Participants) | 58
Age Continuous [Mean (Standard Deviation); unit: Years] | 68.6 (9.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 58
Region of Enrollment [Number; unit: Participants]
  United Kingdom | 4
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Prostate Specific Antigen (PSA) Response
Description: The PSA response was evaluated according to Prostate-Specific Antigen Working Group (PSAWG) criterion, which is, greater than or equal to 50 percent decrease in PSA from Baseline during the study, which would be subsequently confirmed by a measurement that is at least 4 or more weeks after initial documentation of PSA response.
Time Frame: Day 1 of each cycle (of 28 days each) up to Cycle 12
Population: Per protocol population defined as participants who had received at least one dose of abiraterone acetate and must had PSA evaluation/tumor assessment at Baseline and at least 1 post-baseline, and had received a minimum of 3 cycles of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abiraterone
Number analyzed (Participants) | 58
percentage of participants | 37.9 [25.5 to 51.6]

2. Secondary Outcome: Prostate-Specific Antigen Based Progression-free Survival (PSA-PFS)
Description: The PSA-PFS is defined as time to first PSA failure (that is, two consecutive increases in PSA of 50 percent and greater than or equal to 5 nanogram per milliliter, as per Prostate-Specific Antigen Working Group [PSAWG] criterion) or death or the start of secondary anti-tumor therapy, whichever occurs first. If a PSA progression or death does not occur, subject will be censored at the last PSA evaluation.
Time Frame: Baseline and Day 1 of each cycle until first documented disease progression or up to 60 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Abiraterone
Number analyzed (Participants) | 58
days | 141 [110 to 200]

3. Secondary Outcome: Radiographic Progression Free Survival (PFS)
Description: The RAD-PFS is defined as the time from randomization to the earliest objective evidence of radiographic progression or death due to any cause. Progression is defined using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.0, as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Baseline, Day 1 of Cycle 4, 7 and 10, and thereafter every third cycle until first documented disease progression or up to 60 months
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Abiraterone
Number analyzed (Participants) | 58
days | 126 [82 to 333]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the interval from the date of the first dose of abiraterone acetate to the date of death.
Time Frame: Every 3 months until death or up to 60 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Abiraterone
Number analyzed (Participants) | 58
days | 492 [373 to 647]

5. Secondary Outcome: Percentage of Participants With Objective Radiographic Response
Description: Percentage of participants with radiographic objective response is defined as the percentage of participants with complete response (CR) or partial response (PR) as best overall response based on reconciled radiographic disease assessment according to RECIST Version 1.0. The CR is disappearance of all lesions. The PR is at least 30 percent decrease in sum of the longest diameter of target lesions or persistence of one or more non-target lesion(s) or/and maintenance of tumor marker level above the normal limits.
Time Frame: as for outcome 3
Population: Per protocol population defined as participants who had received at least 1 dose of abiraterone acetate and must had PSA evaluation/tumor assessment at Baseline and at least 1 post-baseline, and had received a minimum of 3 cycles of study treatment. "N" (number of participants analyzed) =participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Abiraterone
Number analyzed (Participants) | 48
percentage of participants
  Complete response (CR) | 0
  Partial Response (PR) | 6.3

6. Secondary Outcome: Time to PSA Progression
Description: The time interval from first dose of abiraterone acetate to the date of PSA progression as defined by the Prostate-Specific Antigen Working Group (PSAWG) criteria. If a PSA progression does not occur, subject will be censored at the last PSA evaluation.
Time Frame: Day 8 of Cycle 1, thereafter Day 1 of each cycle up to end of study (60 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Abiraterone
Number analyzed (Participants) | 58
days | 169 [99 to 225]

7. Secondary Outcome: Time to Radiographic Progression
Description: Time to radiographic progression is defined as the time from first dose until the first radiographic progression date that was confirmed.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Abiraterone
Number analyzed (Participants) | 58
days | 88 [82 to 333]

8. Secondary Outcome: Shift From Baseline in Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status Score
Description: ECOG performance status score ranges from 0 to 5 where 0=fully active, perform all pre-disease activities without restriction. 1=restricted in physically strenuous activity but ambulatory, carry out work of a light or sedentary nature, 2=ambulatory, capable of self-care, unable to carry out any work activities, up and about more than (>) 50 percent of waking hours, 3=capable of limited self-care, confined to bed or chair >50 percent of waking hours, 4=completely disabled, not capable of any self-care, totally confined to bed or chair and 5=dead.
Time Frame: Baseline and Day 1 of each cycle until first documented disease progression or up to 60 months
Population: Per protocol population defined as participants who had received at least one dose of abiraterone acetate and must had PSA evaluation/tumor assessment at Baseline and at least 1 post-baseline, and had received a minimum of 3 cycles of study treatment. 'N' (number of participants analyzed) = participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Abiraterone
Number analyzed (Participants) | 57
participants
  Baseline:0; Best Post-dose:0 | 22
  Baseline:0; Best Post-dose:1 | 2
  Baseline:0; Best Post-dose:2 | 0
  Baseline:0; Best Post-dose:3 | 0
  Baseline:0; Best Post-dose:4 | 0
  Baseline:1; Best Post-dose:0 | 14
  Baseline:1; Best Post-dose:1 | 15
  Baseline:1; Best Post-dose:2 | 2
  Baseline:1; Best Post-dose:3 | 0
  Baseline:1; Best Post-dose:4 | 0
  Baseline:2; Best Post-dose:0 | 1
  Baseline:2; Best Post-dose:1 | 1
  Baseline:2; Best Post-dose:2 | 0
  Baseline:2; Best Post-dose:3 | 0
  Baseline:2; Best Post-dose:4 | 0
  Baseline:0; Worst Post-dose:0 | 6
  Baseline:0; Worst Post-dose:1 | 17
  Baseline:0; Worst Post-dose:2 | 1
  Baseline:0; Worst Post-dose:3 | 0
  Baseline:0; Worst Post-dose:4 | 0
  Baseline:1; Worst Post-dose:0 | 0
  Baseline:1; Worst Post-dose:1 | 24
  Baseline:1; Worst Post-dose:2 | 6
  Baseline:1; Worst Post-dose:3 | 1
  Baseline:1; Worst Post-dose:4 | 0
  Baseline:2; Worst Post-dose:0 | 0
  Baseline:2; Worst Post-dose:1 | 0
  Baseline:2; Worst Post-dose:2 | 2
  Baseline:2; Worst Post-dose:3 | 0
  Baseline:2; Worst Post-dose:4 | 0

9. Secondary Outcome: Percentage of Participants With Clinical Benefit
Description: Clinical benefit was defined as an observation of at least 1 of the following: PSA response by PSAWG criteria; radiographic response by RECIST criteria; stable disease by RECIST criteria lasting 6 months; or improvement by at least 1 unit in ECOG performance status.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Abiraterone
Number analyzed (Participants) | 58
percentage of participants
  Disease Stabilization | 12
  Change in participant ECOG score | 16

ADVERSE EVENTS:
Time Frame: Day 8 of Cycle 1 up to End of Study
Arm/Group | Abiraterone
Serious Adverse Events (participants affected / at risk) | 23/58
Other Adverse Events (participants affected / at risk) | 57/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone (N=58)
Anaemia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 1
Fatigue (General disorders) | 2
Pyrexia (General disorders) | 4
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sternal fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood amylase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood potassium increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 2
White blood cell count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 2
Spinal cord compression (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Haematuria (Renal and urinary disorders) | 2
Haemorrhage urinary tract (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Pelvic pain (Reproductive system and breast disorders) | 1
Scrotal swelling (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Aortic stenosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone (N=58)
Anaemia (Blood and lymphatic system disorders) | 15
Lymphopenia (Blood and lymphatic system disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 15
Diarrhoea (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 9
Fatigue (General disorders) | 23
Oedema peripheral (General disorders) | 18
Pain (General disorders) | 4
Pyrexia (General disorders) | 9
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 6
Alanine aminotransferase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 15
Blood albumin decreased (Investigations) | 12
Blood alkaline phosphatase increased (Investigations) | 4
Weight decreased (Investigations) | 10
Anorexia (Metabolism and nutrition disorders) | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 12
Hyperkalaemia (Metabolism and nutrition disorders) | 7
Hypoglycaemia (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 13
Back pain (Musculoskeletal and connective tissue disorders) | 15
Bone pain (Musculoskeletal and connective tissue disorders) | 7
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Headache (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 9
Anxiety (Psychiatric disorders) | 4
Depressed mood (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 4
Dysuria (Renal and urinary disorders) | 4
Haemorrhage urinary tract (Renal and urinary disorders) | 5
Micturition urgency (Renal and urinary disorders) | 3
Nocturia (Renal and urinary disorders) | 4
Pollakiuria (Renal and urinary disorders) | 4
Urinary incontinence (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 4
Hot flush (Vascular disorders) | 6
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less